CLINICAL TRIAL: NCT06448117
Title: Mind Nutrition Study. Effectiveness of Improving Nutrition on Depressive Symptoms and Work Ability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satakunta University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30102023
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depressive Symptoms; Nutrition, Healthy; Quality of Life; Eating Behavior; Work-Related Condition
Keywords: Depressive Symptoms; Nutrient intake; Work ability; Quality of Life; Randomized, controlled trial; Nutritional counseling
MeSH Terms: conditions — Depression; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Subjects in the intervention group participate in a 6-month nutrition counseling program, including two individual and three group-based sessions. The content of the sessions is described in the "Arms and Interventions" section. The behavioral intervention utilizes theoretical frameworks of goal attainment, psychoeducation, peer support, motivational interviewing, mindfulness, and flexible eating restraint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Mind Nutrition" Nutritional counseling (Experimental): The intervention arm includes five dietary counseling sessions during 6 months.
  Interventions: Behavioral: Mind Nutrition
- Control (No Intervention): The control arm does not include any intervention.

INTERVENTIONS:
Behavioral: Mind Nutrition — The 6-month nutrition intervention includes two individual and three group dietary counseling sessions. During the first individual meeting, a research dietitian will assess the participants' diet quality and eating habits, and each participant will set personal goals in cooperation with the research dietitian. At the second individual meeting, the attainment of the goals will be evaluated, and potential challenges and solutions discussed. Each group session has its theme and content in the following chronological order:
  1. Introduction to the theme and importance of a regular meal frequency
  2. Principals of health-promoting diet, mindful eating
  3. Successful eating regulation skills, psychology of the long-term lifestyle changes.
  Additionally, participants receive home assignments and a workbook containing informational material and exercises.
  Arms: "Mind Nutrition" Nutritional counseling

SUMMARY:
The goal of this randomized, controlled trial is to examine the effectiveness of dietary counseling on depressive symptoms, work ability, and quality of life in mental health and substance abuse professionals. The main questions it aims to answer are:

* Whether dietary counseling can lower depressive symptoms and depressive symptoms-related sick leave days and improve work ability among mental health and substance abuse professionals
* Whether dietary counseling can improve life quality, diet quality, and eating behavior among mental health and substance abuse professionals.

Subjects of the intervention group will participate in five dietary counseling sessions during six months. Participants in the control group do not receive any intervention.

Researchers will compare the intervention and control groups to see if dietary counseling is effective in reducing the risk of depressiveness and depression-related sick leave days and improving work ability, quality of life, and nutritional habits.

DETAILED DESCRIPTION:
Background. Depressive disorders are a growing public health concern. Depression is linked to increases in work absenteeism, short-term disability, decreased productivity, and presenteeism and has become a global public health challenge. The association between nutrition and the risk of depressiveness is recognized, but there are no published randomized, controlled whole-diet intervention studies with the main aim of depression prevention. It is essential to investigate the impact of nutrition counseling on symptoms of depression in high-risk groups.

Aims. This Mind Nutrition randomized, controlled trial is part of the Mind Nutrition study that combines the intervention part and a cross-sectional examination that utilizes a separate dataset. The primary aim of the intervention study is to examine whether improving nutrition can (cost-effectively) reduce depressive symptoms and related sick leave and enhance work ability. Secondary aims are to measure the effects of the intervention on diet quality, life quality, and eating behavior, evaluate the attainment of participants' personal goals, and assess the acceptability of the intervention.

Methods. The randomized, controlled trial examines the effectiveness of six-month nutritional counseling on depressive symptoms and work ability among practical and registered nurses and social welfare professionals (n=125) working in the mental health and substance abuse field of the Satakunta wellbeing services county. Half of the participants are randomized into the intervention group and half into the control group. The six-month intervention includes two individual and three group counseling sessions. The control group will not receive any intervention but, instead, continue their habitual diet. The investigators measure the outcomes utilizing questionnaires and three-day food records at baseline and the end of the intervention. Weight and blood pressure will be measured at the same time points.

Discussion. This study will provide nationally and internationally crucial evidence on the effectiveness of nutrition counseling on depressive symptoms, work ability, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 year
* Adequate Finnish language skills
* Work-capable
* Currently employed by Satakunta wellbeing services county for at least 6 months
* Works in the field of mental health and substance abuse
* Education either practical nurse, registered nurse, mental health nurse, or Bachelor of Social Services (in Finnish: Sosionomi)
* Agrees to commit to either of the groups (intervention/control) for 6 months
* Able to give informed consent.

Exclusion Criteria:

* Acute mental health symptoms and incapable to work
* Terminal phase disease or unstable severe chronic disease (consultation of the doctor in charge)
* Employed for a shorter period than 6 months
* Has a history of an eating disorder (consultation of the doctor in charge)
* Center for Epidemiological Studies - Depression (CES-D) score ≥16 and reduced work capacity (presenteeism) (consultation of the medical expert in mental health)
* Substance abuse based on the AUDIT-C score (consultation of the doctor in charge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | 6 months
  Change in depressive symptoms measured with the Center for Epidemiological Studies - Depression (CES-D) questionnaire. It has 20 questions with response options from 0 to 3 points. Possible scores are between 0-60 with higher scores meaning more severe depression symptomology.
Change in work ability | 6 months
  Change in work ability measured with a three-step work ability indicator created by the Finnish Institute for Health and Welfare: "Regardless of whether you are employed or not, please estimate your current work ability." The answer options are coded in three different categories: 1) completely fit for work (2 points), 2) partially unable to work (1 point), and 3) completely unable to work (0 points)."
Change in depressive symptoms-related sick leave days | 6 months
  Change in the number of depressive symptoms-related sick leave days assessed with a structured question.

SECONDARY OUTCOMES:
Change in quality of life | 6 months
  Change in quality of life measured with the World Health Organization Eurohis-QOL (WHO8-EUROHIS) questionnaire. It has eight items with a 5-point response format on a Likert scale. The total score is obtained by summing the eight items and dividing the result by eight, meaning that the possible scores are between 1-5. Higher scores indicate better life quality.
Change in dietary habits | 6 months
  Change in dietary habits assessed with a 163-item Food frequency questionnaire (FFQ) created by the University of Eastern Finland and the Baltic Sea Diet Score derived from the FFQ data. The FFQ comprises nine frequency response options which are multiplied by the portion sizes (grams) to obtain consumption of each listed food item. Average daily food, nutrient, and energy intakes are calculated using the Finnish National Food Composition (Fineli®) database. The Finnish Healthy Diet Index (HDI) score will be derived from the data. Scores range from 0 to 100, with higher scores meaning better diet quality.
Change in energy and nutrient intake | 6 months
  Change in energy and nutrient intake measured with three-day food records utilizing the Eat@Work mobile application by the Satakunta University of Applied Sciences.
Change in eating behavior | 6 months
  Change in Eating behavior assessed by the Three Factor Eating Questionnaire - 18 (TFEQ-18). Its three domains (emotional eating, uncontrolled eating, and cognitive restraint) are measured with 18 questions. Raw scores are scaled to 0-100 points, with higher scores meaning a stronger tendency for each behavior domain.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Kunvik, PhD, Principal Investigator — Senior Researcher
Locations (1):
- Satakunta University of Applied Sciences, Pori, Satakunta, Finland

IPD SHARING:
Plan to Share IPD: No